CLINICAL TRIAL: NCT04158934
Title: Evaluation of Long-term Safety of ADYNOVI/ADYNOVATE (Antihaemophilic Factor [Recombinant] PEGylated, Rurioctocog Alfa Pegol) in Patients With Haemophilia A - An ADYNOVI/ADYNOVATE Post-Authorisation Safety Study (PASS)
Brief Title: A Long-term Study of ADYNOVI/ADYNOVATE in Participants With Haemophilia A
Status: Active, not recruiting | Type: Observational
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: TAK-660-403; EUPAS35698 (Registry Identifier: EUPAS)
Record Dates: First submitted 2019-10-14; First posted 2019-11-12 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — BAX 855; Factor VIII

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Haemophilia A Group: Participants with haemophilia A in the study will receive ADYNOVI/ADYNOVATE prescribed prophylactically by physicians based on their standard clinical practice and in accordance with the national summary of product characteristics (SmPC).
  Interventions: Biological: ADYNOVI/ADYNOVATE

INTERVENTIONS:
Biological: ADYNOVI/ADYNOVATE — Participants will receive ADYNOVI/ADYNOVATE prescribed prophylactically by physicians based on their standard clinical practice and in accordance with the national SmPC.
  Other Names: Antihaemophilic Factor [Recombinant] PEGylated rurioctocog alfa pegol; TAK-660; BAX 855

SUMMARY:
The main aim of this study is to check for long-term side effects from ADYNOVI/ADYNOVATE prophylaxis in participants with haemophilia A when used under standard clinical practice in the real-world clinical setting.

ELIGIBILITY:
Inclusion Criteria

* Signed informed consent obtained from participant and/or legally authorised representative before any study related activities (any procedure related to recording of data according to the protocol).
* Participant at any age with haemophilia A prescribed ADYNOVI/ADYNOVATE prophylaxis.
* Negative factor VIII (FVIII) inhibitor test at study entry.
* Decision to initiate treatment with commercially available ADYNOVI/ADYNOVATE has been made by the participant and/or legally authorised representative and the treating physician before and independently from the decision to include the participant in this study.

Exclusion Criteria

* Previous participation in this study. Participation is defined as signed informed consent.
* Known or suspected hypersensitivity to ADYNOVI/ADYNOVATE or related products.
* Mental incapacity, unwillingness or other barriers precluding adequate understanding or cooperation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 200 participants with haemophilia A will be enrolled. The study will be conducted in European, North American and Asian countries.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2030-02-28 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE) | Throughout the study period (approximately up to 10 years)
  An SAE is any untoward medical occurrence (whether considered to be related to study product or not) that at any dose results in death, life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital abnormality or birth defect, an important medical event. An AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical (study) product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (study) product, whether or not related to the medicinal (study) product. AEs and SAEs that are at least possibly related to study drug ADYNOVI/ADYNOVATE will be evaluated in this outcome.
Number of Participants With Adverse Events of Special Interest (AESI) | Throughout the study period (approximately up to 10 years)
  Adverse events of special interest are as follows: thromboembolic events, hypersensitivity reactions, lack of efficacy and confirmed FVIII inhibitor development.
Number of Participants With Adverse Events (AE) Related to Impaired Renal Function | Throughout the study period (approximately up to 10 years)
  An AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical (study) product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (study) product, whether or not related to the medicinal (study) product. AEs (at least possibly related) that are potentially indicative of or related to long-term effects of PEG accumulation impaired renal function will be evaluated in this outcome.
Number of Participants With Adverse Events (AE) Related to Impaired Hepatic Function | Throughout the study period (approximately up to 10 years)
  An AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical (study) product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (study) product, whether or not related to the medicinal (study) product. AEs (at least possibly related) that are potentially indicative of or related to long-term effects of PEG accumulation impaired hepatic function will be evaluated in this outcome.
Number of Participants With Adverse Events (AE) Related to Impaired Neurologic Function | Throughout the study period (approximately up to 10 years)
  An AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical (study) product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (study) product, whether or not related to the medicinal (study) product. AEs (at least possibly related) that are potentially indicative of or related to long-term effects of PEG accumulation impaired neurologic function will be evaluated in this outcome.

SECONDARY OUTCOMES:
Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Specified Time Points | Baseline, Year 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10
  eGFR levels will be assessed from baseline to end of the study at every visit. Note: all assessments are being done as per Standard of Care (SOC) at each study site/ center and are not mandatory.
Change From Baseline in Alanine Aminotransferase (ALT) at Specified Time Points | Baseline, Year 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10
  ALT levels will be assessed from baseline to end of the study at every visit. Note: all assessments are being done as per Standard of Care (SOC) at each study site/ center and are not mandatory.
Change From Baseline in Bilirubin at Specified Time Points | Baseline, Year 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10
  Bilirubin levels will be assessed from baseline to end of the study at every visit. Note: all assessments are being done as per Standard of Care (SOC) at each study site/ center and are not mandatory.
Change From Baseline in Polyethylene Glycol (PEG) Plasma Levels at Specified Time Points | Baseline, Year 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10
  PEG plasma levels will be assessed from baseline to end of the study at every visit. Note: all assessments are being done as per Standard of Care (SOC) at each study site/ center and are not mandatory.
Number of Participants With Clinically Significant Abnormalities in Vital Signs | Throughout the study period (approximately up to 10 years)
  Clinically significant abnormal findings in vital signs, collected as part of standard of care (SOC)/ standard clinical practice.
Number of Participants With Clinically Significant Abnormalities in Physical Exam | Throughout the study period (approximately up to 10 years)
  Clinically significant abnormal findings in physical exam collected as part of standard of care (SOC)/ standard clinical practice.
Number of Participants With Clinically Significant Abnormalities in Neurological Exam | Throughout the study period (approximately up to 10 years)
  Clinically significant abnormal findings in neurological exam collected as part of standard of care (SOC)/ standard clinical practice.
Number of Participants With Clinically Significant Abnormalities in Clinical Laboratory Parameters | Throughout the study period (approximately up to 10 years)
  Clinically significant abnormal findings in clinical laboratory parameters collected as part of standard of care (SOC)/ standard clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (36):
- UF Health Shands Hospital, Gainesville, Florida, United States
- SHAT of Oncohaematology Diseases, Sofia, Bulgaria
- Croatia (2):
  - Clinical Hospital Sveti Duh, Zagreb
  - University hospital centre Zagreb, Zagreb
- Czechia (2):
  - Fakultni nemocnice v Motole, Prague
  - Krajska zdravotni a.s. - Masarykova nemocnice v Usti nad Labem o.z., Ústí nad Labem
- Germany (4):
  - SRH Kurpfalzkrankenhaus Heidelberg GmbH, Heidelberg, Baden-Wurttemberg
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Universitaetsklinikum Bonn AoeR, Bonn
  - Werlhof-Institut GmbH, Hanover
- Hungary (6):
  - Heim Pal Orszagos Gyermekgyogyaszati Intezet, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Debreceni Egyetem, Debrecen
  - Mohacsi Korhaz, Mohács
  - SzSzB Megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
- Italy (4):
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Azienda Ospedaliera Universitaria Policlinico Umberto I - Università di Roma La Sapienza, Roma
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Torino
- University Medical Centre Groningen-UMCG, Groningen, Netherlands
- South Korea (2):
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (5):
  - Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario de Gran Canaria Dr. Negrin, Las Palmas
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
- Sahlgrenska Universitetssjukhuset, Gothenburg, Sweden
- Taiwan (3):
  - MacKay Memorial Hospital_Tamsui Branch, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District
- Thailand (4):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Phramongkutklao Hospital, Bangkok
  - Siriraj Hospital, Bangkoknoi Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b600d4db2bf003ab48ce6